CLINICAL TRIAL: NCT05516511
Title: Serum Levels of Angiotensin Converting Enzyme in Systemic Lupus Erythematous Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Yasmin Abdelfattah Mohamed, resident doctor at Physical medicine,Rheumatolgy and Rehabilitaion Department , Faculty of medicine, Sohag University, Sohag University
Other Study IDs: Soh-Med-22-08-01
Record Dates: First submitted 2022-08-24; First posted 2022-08-25 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: systemic lupus erythematosus patients
  Interventions: Diagnostic Test: Angiotensin Converting Enzyme test
- control: healthy individuals
  Interventions: Diagnostic Test: Angiotensin Converting Enzyme test

INTERVENTIONS:
Diagnostic Test: Angiotensin Converting Enzyme test — blood sample is taken SLE patients , healthy control , ACE level will be measured by ELISA kits

SUMMARY:
Systemic lupus erythematosus (SLE) is a heterogeneous autoimmune disease that involve many different organs and display a variable clinical course.The prevalence of SLE varies across gender, race/ethnicity, and geographic regions. SLE demonstrates a striking female predominance with a peak incidence of disease during the reproductive years. In adults, the female to male ratio is 10- Renal involvement is common in SLE and is a significant cause of morbidity and mortality. It is estimated that as many as 90% of patients with SLE will have pathologic evidence of renal involvement on biopsy, but clinically significant nephritis will develop in only 50%. AII is a potent pro-inflammatory modulator with the ability to augment the immune responses in renal and non-renal tissues. Specifically in the kidney, AII stimulates mononuclear cells, favoring hyperplasia and hypertrophy of mesangial, tubular cells and interstitial fibroblasts, and increases expression and synthesis of the extracellular protein matrix leading to fibrosis.

Angiotensin II and strong candidate for a mediator of the development and progression of renal disease in SLE has been found to promote glomerular cell proliferation, alter growth factor expression, and activate proinflammatory cytokines, all of which promote glomerulosclerosis

ELIGIBILITY:
Inclusion Criteria:

* 1-Patients who fulfill the 2019 American College of Rheumatology/European League against Rheumatism classification criteria of Systemic Lupus Erythematosus 2-Patients diagnosed as lupus nephritis , actually did renal biobsy 3-Patients who is able to give informed consent to join the study

Exclusion Criteria:

* - Any patient with any collagen disease other than systemic lupus erythematosus.

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will include 50 patients diagnosed by 2019 American College of Rheumatology/European League Against Rheumatism classification criteria as systemic lupus erythematosus, 25of them will be selected as Lupus Nephritis (LN).
  - 25 normal healthy persons matched for age and sex as control group.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Angiotensin Converting Enzyme test | 3 months
  laboratory test, ELISA kits, measure serum levels of angiotensin converting enzyme in SLE patients , control
protein creatine ratio | 3 months
  laboratory test, urine sample used to measure amount of proteinurea
serum creatine test | 3 months
  lab test , to asses renal function

SECONDARY OUTCOMES:
Anti nuclear Anti body tset | 3 months
  lab tset, IF technique, for diagnosis of SLE disease
anti ds-DNA test | 3 months
  lab test , for diagnosis of SLE , lupus nephritis

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Pons-Estel GJ, Alarcon GS, Scofield L, Reinlib L, Cooper GS. Understanding the epidemiology and progression of systemic lupus erythematosus. Semin Arthritis Rheum. 2010 Feb;39(4):257-68. doi: 10.1016/j.semarthrit.2008.10.007. Epub 2009 Jan 10. PMID 19136143
- [Background] Weening JJ, D'Agati VD, Schwartz MM, Seshan SV, Alpers CE, Appel GB, Balow JE, Bruijn JA, Cook T, Ferrario F, Fogo AB, Ginzler EM, Hebert L, Hill G, Hill P, Jennette JC, Kong NC, Lesavre P, Lockshin M, Looi LM, Makino H, Moura LA, Nagata M; International Society of Nephrology Working Group on the Classification of Lupus Nephritis; Renal Pathology Society Working Group on the Classification of Lupus Nephritis. The classification of glomerulonephritis in systemic lupus erythematosus revisited. Kidney Int. 2004 Feb;65(2):521-30. doi: 10.1111/j.1523-1755.2004.00443.x. PMID 14717922
- [Background] Ruiz-Ortega M, Ruperez M, Esteban V, Rodriguez-Vita J, Sanchez-Lopez E, Carvajal G, Egido J. Angiotensin II: a key factor in the inflammatory and fibrotic response in kidney diseases. Nephrol Dial Transplant. 2006 Jan;21(1):16-20. doi: 10.1093/ndt/gfi265. Epub 2005 Nov 9. PMID 16280370
- [Background] Klahr S, Morrissey JJ. The role of vasoactive compounds, growth factors and cytokines in the progression of renal disease. Kidney Int Suppl. 2000 Apr;75:S7-14. PMID 10828755